CLINICAL TRIAL: NCT06646991
Title: Comparison of Several Oxygenation Targets With Different Oxygen Interfaces - Impact on Oxygen Flow Rates
Acronym: Interfaces
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, François Lellouche, Principal Investigator, Laval University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-4198
Record Dates: First submitted 2024-06-17; First posted 2024-10-17 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Oxygen Toxicity; COPD Bronchitis; Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nellcor oximeter (Other)
  Interventions: Device: Nasal canula - up to 6 liters per minute; Device: Nasal canula - up to 15 liters per minute; Device: Open oxygen mask; Device: Simple oxygen face mask
- Nonin Oximeter (Other)
  Interventions: Device: Nasal canula - up to 6 liters per minute

INTERVENTIONS:
Device: Nasal canula - up to 6 liters per minute — Oxygen will be administered via nasal cannula up to 6 liters per minute during this period.
  Oxygen flow rates will be adjusted manually, with a gradual increase in flow rates to achieve a oxygen flow rates for reach the peripheral oxygen saturation (SpO2) target (92% for non chronic obstructive pulmonary disease (non COPD) patient and 90% for chronic obstructive pulmonary disease (COPD) patient).
  The steady state will be defined by a fixed oxygen flow rate and a stable SpO2 around the target ±2% for 15 minutes. The average oxygen flow rate during the last five minutes will be used.
Device: Nasal canula - up to 15 liters per minute — Oxygen will be administered via nasal cannula up to 15 liters per minute during this period.
  Oxygen flow rates will be adjusted manually, with a gradual increase in flow rates to achieve a oxygen flow rates for reach the SpO2 target (92% for non COPD patient and 90% for COPD patient).
  The steady state will be defined by a fixed oxygen flow rate and a stable SpO2 around the target ±2% for 15 minutes. The average oxygen flow rate during the last five minutes will be used.
  Arms: Nellcor oximeter
Device: Open oxygen mask — Oxygen will be administered via an open during this period. Oxygen flow rates will be adjusted manually, with a gradual increase in flow rates to achieve a oxygen flow rates for reach the SpO2 target (92% for non COPD patient and 90% for COPD patient).
  The steady state will be defined by a fixed oxygen flow rate and a stable SpO2 around the target ±2% for 15 minutes. The average oxygen flow rate during the last five minutes will be used.
  Arms: Nellcor oximeter
Device: Simple oxygen face mask — Oxygen will be administered via simple oxygen face mask during this period. Oxygen flow rates will be adjusted manually, with a gradual increase in flow rates to achieve a oxygen flow rates for reach the SpO2 target (92% for non COPD patient and 90% for COPD patient).
  The steady state will be defined by a fixed oxygen flow rate and a stable SpO2 around the target ±2% for 15 minutes. The average oxygen flow rate during the last five minutes will be used.
  Arms: Nellcor oximeter

SUMMARY:
Oxygen therapy is at the heart of the healthcare system. Oxygen flow rates depend on a number of confounding factors confounding factors (target used, skin pigmentation, pulse oximeter used, etc.) The investigators have recently have recently demonstrated that the combination of these factors (different peripheral oxygen saturation (SpO2) targets and different oximeters) can have a significant impact on oxygen flows rates. The effect on oxygen flow was not simply additive .

The aim of this study is to evaluate the impact of the interface used on oxygen flow rates in different patient populations (main objective). The investigatoers also evaluate the impact of the interface on carbon dioxide (PaCO2), in particular with closed oxygen masks, with which rebreathing is theoretically possible (secondary objective).

secondary objective).

ELIGIBILITY:
Inclusion Criteria:

* Adult (> or = 18 years old)
* Ongoing on conventional oxygen therapy with peripheral oxygen saturation (SpO2) between 88 and 100% with the usual oximeter
* SpO2 < 92% ambient air with the usual oximeter

Exclusion Criteria:

* No SpO2 signal with with the usual oximeter
* False nails or nail polish
* Severe anemia documented on last blood count during current hospitalization (haemoglobin (Hb) < 80g/L)
* Oxygen flow > 6 L/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Oxygen flow | Mean Oxygen flow in the five last minute of each study period (between minute 10 and 15)
  Oxygen flows (or fraction of inspired oxygen (FiO2)) at the end of each study period (last minute average) to reach peripheral oxygen saturation (SpO2) target to reach SpO2 target with specific oxygen administration interfaces

SECONDARY OUTCOMES:
Partial oxygen weaning | Mean oxygen flow in the five last minute of each study period (between minute 10 and 15)
  Rate of partial oxygen weaning (Oxygen flow <=0.5 L/min)
Complete oxygen weaning | Mean oxygen flow in the five last minute of each study period (between minute 10 and 15)
  Rate of complete oxygen weaning (Oxygen flow =0 L/min or FiO2 0.21)

OTHER OUTCOMES:
Gaps between the different oximeters | through period completion, minute 15
  Average of the SpO2 value gaps between the different oximeters tested
Gaps between PaCO2 | through period completion, minute 15
  PaCO2 value at the end of the period

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Canada

IPD SHARING:
Plan to Share IPD: No